CLINICAL TRIAL: NCT07181382
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Oral Inhalation of Seralutinib for the Treatment of Pulmonary Hypertension Associated With Interstitial Lung Disease (PH-ILD) Followed by a Long-Term Extension Evaluating Safety and Efficacy
Brief Title: Efficacy and Safety of Seralutinib in Adult Subjects With Pulmonary Hypertension Associated With Interstitial Lung Disease (PH-ILD)
Acronym: SERANATA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: GB002, Inc. (Industry)
Collaborators: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Organization: Gossamer Bio Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GB002-3201; 2025-521777-13-00 (EU CTIS Number)
Record Dates: First submitted 2025-09-12; First posted 2025-09-18 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Pulmonary Hypertension Associated With Interstitial Lung Disease
Keywords: seralutinib; GB002; SERANATA; Pulmonary hypertension; Interstitial lung disease
MeSH Terms: conditions — Hypertension, Pulmonary; Lung Diseases, Interstitial

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo inhaled orally twice daily (BID) for 24 weeks in PCP. Subjects randomized to the placebo treatment group in the PCP will receive seralutinib in LTE.
  Interventions: Drug: Placebo; Drug: Seralutinib; Device: Generic Dry Powder Inhaler
- Seralutinib 90 mg (Experimental): Seralutinib inhaled orally BID for 24 weeks in PCP. Seralutinib inhaled orally BID up to 144 weeks in LTE.
  Interventions: Drug: Seralutinib; Device: Generic Dry Powder Inhaler
- Seralutinib 120 mg (Experimental): Seralutinib inhaled orally BID for 24 weeks in PCP. Seralutinib inhaled orally BID up to 144 weeks in LTE.
  Interventions: Drug: Seralutinib; Device: Generic Dry Powder Inhaler

INTERVENTIONS:
Drug: Placebo — Matching capsule containing placebo
  Arms: Placebo
Drug: Seralutinib — Capsule containing seralutinib
Device: Generic Dry Powder Inhaler — Generic dry powder inhaler for seralutinib or placebo delivery

SUMMARY:
This Phase 3 study is designed as a 24-week randomized, double-blind, placebo-controlled period (PCP) followed by a 144-week long-term extension (LTE) period. The primary objective of the PCP is to evaluate the effect of seralutinib on improving exercise capacity in subjects with World Health Organization (WHO) Group 3 pulmonary hypertension associated with interstitial lung disease. The primary objective of the LTE is to evaluate the long-term safety and tolerability of seralutinib.

ELIGIBILITY:
Inclusion Criteria:

1. Adult subjects aged 18 years to 80 years, inclusive, at the time of voluntarily signing the informed consent form, prior to initiation of any study-specific activities/procedures.
2. Body mass index (BMI) ≥ 15 kg/m2 and ≤ 40 kg/m2.
3. A diagnosis of WHO Group 3 pulmonary hypertension (PH) associated with interstitial lung disease.
4. Right heart catheterization at Screening meeting the following criteria:

   1. Pulmonary vascular resistance (PVR) ≥ 4 Woods Units, AND
   2. Pulmonary capillary wedge pressure (PCWP) or left ventricular end diastolic pressure (LVEDP) ≤ 15 mm Hg, AND
   3. Mean pulmonary arterial pressure (mPAP) ≥ 25 mm Hg. Historic RHC up to 12 weeks prior to Screening may be acceptable for eligibility.
5. Forced vital capacity (FVC) ≥ 45% predicted at Screening.
6. Screening 6MWD of ≥ 100 m and ≤ 475 m.
7. Subjects receiving permitted chronic medication for underlying fibrotic ILD must be receiving background therapy from at least 16 weeks prior to Screening.
8. Subjects receiving SARD medication must be receiving background therapy from at least 16 weeks prior to Screening.
9. Subjects on supportive medications (eg, diuretics) must be on an optimized dose for ≥ 30 days prior to and throughout Screening.
10. In the opinion of the Investigator, the subject has no other medical conditions that impair the proper use of the inhaler.
11. Women of childbearing potential (WOCBP) must have a negative serum pregnancy test at Screening and a negative urine pregnancy test on PCP Day 1 before first administration of IP.
12. WOCBP who are not abstinent and intend to be sexually active with a non-sterilized male partner must be willing to use a highly effective method of contraception from consent through 30 days following the last administration of IP.
13. Women of nonchildbearing potential (WONCBP), classified by 1 of the following:

    1. Surgical sterilization
    2. Evidence of post-menopausal status.
14. Male subjects: Non-sterilized male subjects who are not abstinent and intend to be sexually active with a female partner of childbearing potential must use a male condom from consent through 90 days after the last dose of IP.

Exclusion Criteria:

1. Diagnosis of pulmonary arterial hypertension (PAH) or PH other than WHO Group 3.
2. PH associated with sarcoidosis, combined pulmonary fibrosis and emphysema, chronic obstructive pulmonary disease, or progressive massive fibrosis.
3. Human immunodeficiency virus (HIV).
4. Uncontrolled atrial fibrillation or paroxysmal atrial fibrillation.
5. History of a potentially life-threatening cardiac arrhythmia with an ongoing risk.
6. Uncontrolled systemic hypertension
7. Subjects receiving > 10 L/min of oxygen supplementation via nasal cannula at rest or > 15 L/min during six-minute walk tests conducted during Screening.
8. Acute pulmonary embolism within 12 weeks prior to and throughout Screening.
9. Untreated moderate or severe obstructive sleep apnea.
10. Clinically significant history of liver disease (ie, Child-Pugh Class A - C, viral hepatitis, liver cirrhosis, hepatobiliary disorders, etc).
11. History of malignancy within 5 years prior to Screening, with the exception of localized and adequately treated non-metastatic basal and squamous cell carcinoma of the skin and in-situ carcinoma of the cervix.
12. Uncontrolled bacterial, viral, or fungal infections which require ongoing systemic therapy.
13. Severe acute or chronic medical or laboratory abnormality that may increase the risk associated with study participation or IP administration, or absolute neutrophil count (ANC) < 1 x 109/L.
14. Pregnant or nursing or intends to become pregnant during the duration of the study.
15. Major surgical procedures planned to occur during trial period.
16. Any other medical condition or laboratory abnormality that, in the opinion of the Investigator, would prohibit the subject from participating in the study, eg, severe concomitant illness limiting life expectancy (< 24 weeks).
17. Body weight < 40 kg at Screening.
18. Estimated glomerular filtration rate (eGFR) < 45 mL/min/1.73 m2
19. Evidence of active Hepatitis B or Hepatitis C, or active tuberculosis (TB) infections at Screening.
20. Subjects receiving both nintedanib and pirfenidone.
21. Initiation of an exercise program for cardiopulmonary rehabilitation within 12 weeks prior to and throughout Screening or planned during their time on the PCP.
22. Prior participation in seralutinib studies and/or prior treatment with seralutinib.
23. Currently participating in or has participated in a study of an investigational agent or has used an investigational device for the treatment of PH-ILD within 12 weeks or 5 half-lives of the investigational agent, whichever is longer, prior to Screening.
24. Current use or within 24 weeks prior to Randomization of inhaled tobacco- or nicotine-containing products (including e-vapor products) and/or inhaled marijuana.
25. Current alcohol use disorder based on the opinion of the Investigator, and/or a positive test for drugs of abuse at Screening.
26. Subjects with a history of severe milk protein allergy.
27. QT interval corrected for heart rate using Fridericia's formula (QTcF) of > 500 msec.
28. In the opinion of the Investigator, the subject has any condition that would interfere with the interpretation of study assessments or has any disease or condition that would likely be the primary limit to ambulation (as opposed to PH).

NOTE: Additional inclusion/exclusion criteria may apply, per protocol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Change in distance achieved on the six-minute walk test (6MWT), from baseline to PCP Week 24 | Baseline to PCP Week 24
Incidence of treatment-emergent adverse events | From first dose of LTE study treatment through LTE Week 148

SECONDARY OUTCOMES:
Time to first event of Adjudication Committee (AC)-confirmed clinical worsening from first dose of investigational product (IP) through PCP Week 24 | Baseline to PCP Week 24
  Event is defined as:
  * Death (all causes)
  * Hospitalization for ≥ 24 hours due to a worsening cardiopulmonary indication
  * ≥ 15% 6MWD decline from baseline, directly related to PH-ILD assessed by two 6MWTs at least 4 hours apart and no more than 1 week apart
Change in N-terminal pro b-type natriuretic peptide (NT-proBNP) from baseline to PCP Week 24 | Baseline to PCP Week 24
Change in absolute forced vital capacity (FVC) from baseline to PCP Week 24 | Baseline to PCP Week 24
Proportion of subjects meeting each AC-confirmed component of clinical worsening by PCP Week 24 | Baseline to PCP Week 24
  Components of clinical worsening are defined for the first secondary outcome measure above.
Change in Euro-QoL - 5 Dimensions - 5 Levels (EQ-5D-5L) from baseline to PCP Week 24 | Baseline to PCP Week 24
  The EQ-5D-5L is a patient questionnaire that includes two components. The first is the EQ-5D-5L descriptive system, which profiles a subject's current health state across 5 dimensions (Mobility, Self-Care, Usual Activities, Pain/Discomfort, Anxiety/Depression). Each dimension is comprised of a single question with 5 possible responses that are scored 1-5, corresponding to no problems, slight problems, moderate problems, severe problems, and unable to/extreme problems, respectively. Higher scores for a dimension mean a worse outcome. The second is a visual analogue scale (EQ VAS), which asks a subject to assess their overall health. The EQ VAS has a range of 0-100, with a higher score representing a better outcome.
Change in Living with Pulmonary Fibrosis (L-PF) from baseline to PCP Week 24 | Baseline to PCP Week 24
Changes in distance achieved on the 6MWT | LTE Week 12 to LTE Week 148
Changes in NT-proBNP | LTE Week 4 to LTE Week 148
Changes in absolute forced vital capacity (FVC) | LTE Week 12 to LTE Week 148

CONTACTS AND LOCATIONS:
Overall Officials: Richard Aranda, MD, Study Director — Gossamer Bio Inc.
Locations (4):
- United States (3):
  - Valley Advanced Lung Diseases Institute, Fresno, California
  - University of New Mexico Health Sciences Center, Albuquerque, New Mexico
  - Pulmonary Associates of Richmond, Inc., Richmond, Virginia
- Hillel Yaffe Medical Center, Hadera, Israel

IPD SHARING:
Plan to Share IPD: No